CLINICAL TRIAL: NCT03968718
Title: PATIENT VOICES - A Project for the Integration of Systematic Assessment of Patient Reported Outcomes Within an E-Health Program in an Italian Comprehensive Cancer Center
Brief Title: PATIENT VOICES Integration of Systematic Assessment of Patient Reported Outcomes Within Clinical Oncology Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Cinzia Brunelli, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Istitutotumori
Record Dates: First submitted 2019-02-05; First posted 2019-05-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Neoplasms; Symptoms and Signs; Psychological Distress; Satisfaction, Consumer; Quality of Life
Keywords: Patient Reported Outcome Measures; Feasibility study
MeSH Terms: conditions — Neoplasms; Signs and Symptoms; Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systematic ePROMs Assessment (Experimental): Intervention: The intervention is constituted by a Systematic ePROMs Assessment in routine cancer care in a comprehensive cancer centre.
  This will involve preliminary sensitization and training of both clinicians and patients towards the use of ePROMs.
  Data filled in by patients through electronic devices will be prompt made available to the clinician during the patient examination.
  Interventions: Behavioral: Systematic ePROMs Assessment

INTERVENTIONS:
Behavioral: Systematic ePROMs Assessment — Depending on the care setting, eligible patients will be asked to fill in one of the following e-PROMs assessment:
  Edmonton symptom assessment scale (ESAS-r) (outpatients)
  Distress Thermometer (inpatients)
  An ad hoc questionnaire adapted from the Bench-Can and EURACAN projects plus the institutional customer satisfaction survey (patients followed by multidisciplinary teams)

SUMMARY:
Listening to "patient voices" in terms of symptoms, emotional status, satisfaction with care and information received, represents a major shift in medicine. It is in fact crucial in medical decision making and patient empowerment, especially in cancer care.

Patient Reported Outcomes Measures (PROMs) and in particular electronically assessed PROMS (ePROMS), have been identified as potentially effective tools to systematically gather patient voices. Despite international extensive and growing interest, systematic PROM collection is not widely implemented in routine cancer care, due to barriers at various levels.

The PATIENT VOICES is a project aimed at achieving a stepwise inclusion and integration of PROMs within routine clinical practice at the FONDAZIONE IRCCS ISTITUTO NAZIONALE TUMORI-MILANO. Phase I of the Patient Voices project (pilot and feasibility testing), will be the focus of the present study and its results will be the base for subsequent phases (implementation and impact assessment).

DETAILED DESCRIPTION:
Study aims of this phase are:

* Assessing the use and attitudes toward PROMs by clinicians in a comprehensive cancer centre.
* Reviewing and compare pre-existing ePROMS assessment systems.
* Developing and pilot testing a flexible system for electronic collection of PROMs.
* Assessing feasibility of ePROM assessment of physical symptoms, psychological distress and patient satisfaction.
* Identifying barriers to and developing strategies for the final implementation and integration of routine ePROMs into the clinical practice.

The project will last 2 years. Longitudinal and cross-sectional studies will be carried out with the aim to evaluate compliance, acceptability, and usability of a routine ePROM assessment system by both patients and clinicians. Participants will be enrolled among patients attending 3 out-patient clinics (physical symptom), 3 inpatient wards (psychological distress) and 5 multidisciplinary teams (patient satisfaction). The Edmonton symptom assessment scale, the Distress Thermometer, and a questionnaire adapted from the Bench-Can and EURACAN projects plus the institutional customer satisfaction survey, will be used in the three studies. Qualitative methods will be used identify patient and clinician related barriers to ePROM assessment and to pinpoint engagement strategies to promote its use in routine cancer care. Semi-structured interviews and focus groups will be carried out.

Quantitative and qualitative studies will respectively enroll 600 and 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* a verified cancer diagnosis

Exclusion Criteria:

* inability to fill in PROMs due to cognitive impairment, psychological disturbance or language problems as judged by the study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient compliant with ePROM assessment | Baseline (one-time point only)
  Compliant patients are defined as patients successfully completing ePROM assessment.
Proportion of clinical encounters using ePROM assessment | Baseline (one-time point only)
  Clinical encounters using ePROM assessment are encounters in which the clinician gets access to symptom or psychological distress data collected by the patients through ePROM assessment

SECONDARY OUTCOMES:
Proportion of patient compliant with ePROM repeated assessments | 6 months
  Proportion patients who succesfully complete ePROMs assessments at each follow-up visit
Proportion of refusals | Baseline (one-time point only)
  Proportion of patients refusing to use the system and reason for refusal

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Brunelli, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunelli C, Alfieri S, Zito E, Spelta M, Arba L, Lombi L, Caselli L, Caraceni A, Borreani C, Roli A, Miceli R, Tine' G, Zecca E, Platania M, Procopio G, Nicolai N, Battaglia L, Lozza L, Shkodra M, Massa G, Loiacono D, Apolone G. Patient Voices: Multimethod Study on the Feasibility of Implementing Electronic Patient-Reported Outcome Measures in a Comprehensive Cancer Center. JMIR Cancer. 2025 Jan 22;11:e56625. doi: 10.2196/56625. PMID 39842002
- [Derived] Brunelli C, Borreani C, Caraceni A, Roli A, Bellazzi M, Lombi L, Zito E, Pellegrini C, Spada P, Kaasa S, Foschi AM, Apolone G; PATIENT VOICES study group. PATIENT VOICES, a project for the integration of the systematic assessment of patient reported outcomes and experiences within a comprehensive cancer center: a protocol for a mixed method feasibility study. Health Qual Life Outcomes. 2020 Jul 28;18(1):252. doi: 10.1186/s12955-020-01501-1. PMID 32723341